CLINICAL TRIAL: NCT03491462
Title: A Phase 3, Randomised, Placebo-Controlled Trial of Arimoclomol in Amyotropic Lateral Sclerosis
Brief Title: Arimoclomol in Amyotropic Lateral Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ZevraDenmark (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORARIALS-01
Record Dates: First submitted 2018-03-27; First posted 2018-04-09 (Actual); Results first posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Arimoclomol; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — arimoclomol

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, parallel group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arimoclomol (Experimental): 248 mg arimoclomol base (equivalent to 400 mg arimoclomol citrate) 3 times daily
  Interventions: Drug: Arimoclomol
- Placebo (Placebo Comparator): 248 mg matching placebo 3 times daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Arimoclomol — 2 capsules (2 x 124 mg arimoclomol base; equivalent to 2 x 200 mg arimoclomol citrate) taken 3 times daily
  Arms: Arimoclomol
Drug: Placebo — 2 matched placebo capsules taken 3 times daily
  Arms: Placebo

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled, parallel group trial to evaluate the efficacy and safety of arimoclomol in amyotropic lateral sclerosis (ALS)

DETAILED DESCRIPTION:
Screening up to 4 weeks Treatment up to 76 weeks

ELIGIBILITY:
Inclusion Criteria:

* Subject meets revised El Escorial criteria for clinically possible, clinically probable / clinically probable ALS laboratory-supported, clinically definite ALS or clinically definite familial ALS laboratory-supported
* 18 months or less since first appearance of weakness (e.g. limb weakness, dysarthria, dysphagia, shortness of breath)
* ALS Functional Rating Scale-Revised (ALSFRS-R) equal to or above 35 and erect (seated) Slow Vital Capacity (SVC) % predicted equal to or above 70% at Screening

Exclusion Criteria:

* Tracheostomy or use of non-invasive ventilation for more than 2 hours during waking hours at the time of Screening and Baseline
* Pregnant or breast-feeding
* Current or anticipated use of diaphragmatic pacing
* Any other relevant medically significant condition which could present risk to the subject or interfere with the assessment of safety or has an increased risk of causing death during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Benatar, MD PhD, Principal Investigator — University of Miami
Locations (29):
- United States (10):
  - St. Joseph's Hospital and Medical Center (SJHMC) - Barrow Neurological Institute (BNI) - The Gregory W. Fulton ALS and Neuromuscular Disease Center, Phoenix, Arizona
  - HonorHealth Neurology, Phoenix, Arizona
  - UC Irvine Health ALS and Neuromuscular Center, Orange, California
  - University of Miami, Miami, Florida
  - University of Kansas Medical Center (KUMC) - Landon Center on Aging, Kansas City, Kansas
  - Hospital for Special Surgery, New York, New York
  - Providence Brain & Spine Institute, Portland, Oregon
  - University of Pensylvania, Perelman Center for Advanced Medicine - Penn Neuroscience Center, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Virginia Health System, Charlottesville, Virginia
- Catholic University Leuven, Leuven, Belgium
- Canada (3):
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- France (2):
  - Centre Hospitalier Regional Universitaire (CHRU) Montpellier - Hopital Gui De Chauliac, Montpellier
  - Groupe Hospitalier Pitie-Salpetriere - Centre d'Investigation Clinique Neurosciences 1422, Paris
- Germany (3):
  - Charite - Universitaetsmedizin Berlin - Campus Virchow-Klinikum (CVK) - Ambulanz fuer ALS und andere Motoneuronenerkrankungen, Berlin
  - Medizinische Hochschule Hannover (MHH) - Klinik fuer Neurologie, Hanover
  - Universitaetsklinikum Ulm - Klinik fuer Neurologie, Ulm
- Italy (2):
  - Instituti Clinica Scientifici Maugeri - IRCCS, Milan
  - Azienda Ospedaliero Universitaria (AUO) di Torino - Citta'della Salute e della Scienza di Torino, Torino
- University Medical Center Utrecht, Utrecht, Netherlands
- Poland (2):
  - Centrum Medyczne NeuroProtect, Warsaw
  - Citi Clinic, Warsaw
- Spain (2):
  - Hospital Universitario Vall d'Hebron ALS Unit. Consultas Externas; Office: 9-10-11, Barcelona
  - Hospital Carlos III - Hospital Universitario La Paz, ALS Unit, Madrid
- Umeå University Hospital, Umeå, Sweden
- Kantonsspital St.Gallen, Muskelzentrum/ALS Clinic, Sankt Gallen, Switzerland
- Leonard Wolfson Experimental Neurology Centre, London, United Kingdom

REFERENCES:
- [Derived] Benatar M, Hansen T, Rom D, Geist MA, Blaettler T, Camu W, Kuzma-Kozakiewicz M, van den Berg LH, Morales RJ, Chio A, Andersen PM, Pradat PF, Lange D, Van Damme P, Mora G, Grudniak M, Elliott M, Petri S, Olney N, Ladha S, Goyal NA, Meyer T, Hanna MG, Quinn C, Genge A, Zinman L, Jabari D, Shoesmith C, Ludolph AC, Neuwirth C, Nations S, Shefner JM, Turner MR, Wuu J, Bennett R, Dang H, Sundgreen C; ORARIALS-01 trial team. Safety and efficacy of arimoclomol in patients with early amyotrophic lateral sclerosis (ORARIALS-01): a randomised, double-blind, placebo-controlled, multicentre, phase 3 trial. Lancet Neurol. 2024 Jul;23(7):687-699. doi: 10.1016/S1474-4422(24)00134-0. Epub 2024 May 20. PMID 38782015

RESULTS

PARTICIPANT FLOW:
Groups:
- Arimoclomol (up to 76 Weeks): Arimoclomol base 248 mg 3 times daily for up to 76 weeks
- Placebo (up to 76 Weeks): Matching placebo 3 times daily for up to 76 weeks
Period: Overall Study
Arm/Group | Arimoclomol (up to 76 Weeks) | Placebo (up to 76 Weeks)
Started | 160 (The 160 participants in the modified intention-to-treat (mITT) population excludes 3 participants in the edaravone sub-population (participants on minimum 6 months' stable treatment with edaravone and who otherwise fulfil the eligibility criteria)) | 79 (The 79 participants in the modified intention-to-treat (mITT) population excludes 3 participants in the edaravone sub-population (participants on minimum 6 months' stable treatment with edaravone and who otherwise fulfil the eligibility criteria))
Completed | 122 (Participants who reached a survival endpoint (PAV / tracheostomy / death) during the study were recorded as completers) | 63 (Participants who reached a survival endpoint (PAV / tracheostomy / death) during the study were recorded as completers)
Not Completed | 38 | 16
Not completed — Lost to Follow-up | 2 | 0
Not completed — Adverse Event | 11 | 1
Not completed — Physician Decision | 3 | 0
Not completed — Withdrawal by Subject | 22 | 15

BASELINE CHARACTERISTICS:
Population: All participants in the modified intention-to-treat (mITT) population
Groups:
- Total: Total of all reporting groups
Arm/Group | Arimoclomol (up to 76 Weeks) | Placebo (up to 76 Weeks) | Total
Number analyzed (Participants) | 160 | 79 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (11.26) | 56.6 (9.97) | 57.6 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 34 | 88
  Male | 106 | 45 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 7 | 20
  Not Hispanic or Latino | 132 | 64 | 196
  Unknown or Not Reported | 15 | 8 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 136 | 66 | 202
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 23 | 11 | 34
Revised ALS Functional Rating Scale (ALSFRS-R) [Mean (Standard Deviation); unit: units on a scale] — The ALSFRS-R score is based on a rating scale where 12 functions are rated on 5-point ordinal rating scales (from 0 to 4) with a maximum score of 48 (sum of all 12 items). The higher the score the better functioning.
  units on a scale | 40.6 (3.93) | 40.2 (3.65) | 40.5 (3.83)
Percent (%) Predicted Slow Vital Capacity (SVC) [Mean (Standard Deviation); unit: percent (%) predicted SVC] — Slow Vital Capacity (SVC) is a measure of breathing function. SVC measures the volume that can be exhaled from a full inhalation after exhaling to a maximum as slowly as possible. The percent (%) of predicted SVC is reported.
  percent (%) predicted SVC | 95.8 (15.98) | 98.1 (14.78) | 96.5 (15.60)

OUTCOME MEASURES:

1. Primary Outcome: Combined Assessment of Function and Survival (CAFS)
Description: Combined Assessment of Function and Survival (CAFS) is a composite endpoint that includes 1) the change from baseline in revised ALS functional rating scale (ALSFRS-R) and 2) the survival endpoint (time to permanent assisted ventilation [PAV], tracheostomy or death).
  On the ALSFRS-R, 12 functions are rated on 5-point ordinal rating scales (from 0 to 4) with a total score range (minimum and maximum score) of 0-48 (sum of all 12 items). The higher the score the better functioning.
  For the survival endpoint, the longer time to PAV, tracheostomy, or death the better outcome.
  A patient's CAFS score represents a patient's rank in the study based on comparing the patient's outcome for both the change in ALSFRS-R and the time to event (PAV, tracheostomy, or death) to the outcome for all other patients in the study in a pairwise fashion. A higher rank score (range 0-1) is considered a better outcome.
  The reported values are the mean rank scores in each group for the composite endpoint.
Time Frame: Over 76 Weeks
Population: modified intention-to-treat (mITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arimoclomol (up to 76 Weeks) | Placebo (up to 76 Weeks)
Number analyzed (Participants) | 160 | 79
score on a scale | 0.51 (0.291) | 0.49 (0.283)
Statistical Analysis 1: Comparison: Arimoclomol (up to 76 Weeks) vs Placebo (up to 76 Weeks); Test type: Superiority; p = 0.6208, Gehan's extended Wilcoxon's test

2. Secondary Outcome: Time to Permanent Assisted Ventilation (PAV) / Tracheostomy / Death
Description: Time from baseline to one of the events (PAV / tracheostomy / death). PAV is defined as the first of 7 consecutive days on which PAV was used for >22 hours/day
Time Frame: Over 76 weeks
Population: modified intention-to-treat (mITT)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Arimoclomol (up to 76 Weeks) | Placebo (up to 76 Weeks)
Number analyzed (Participants) | 160 | 79
days | NA [479 to NA] — Median and 3rd Quartile was not estimable due to an insufficient number of participants with events | NA [466 to NA] — Median and 3rd Quartile was not estimable due to an insufficient number of participants with events

3. Secondary Outcome: Change From Baseline to Week 76 (or End-of-trial) in the Revised ALS Functional Rating Scale (ALSFRS-R)
Description: The ALSFRS-R score is based on a rating scale where 12 functions are rated on 5-point ordinal rating scales (from 0 to 4) with a maximum score of 48 (sum of all 12 items). The higher the score the better functioning.
Time Frame: Week 76 (or end of trial)
Population: modified intention-to-treat (mITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arimoclomol (up to 76 Weeks) | Placebo (up to 76 Weeks)
Number analyzed (Participants) | 160 | 79
units on a scale | -15.4 (8.71) | -15.0 (9.10)

4. Secondary Outcome: Change From Baseline to Week 76 (or End-of-trial) in Percent (%) Predicted Slow Vital Capacity (SVC)
Description: Slow Vital Capacity (SVC) is a measure of breathing function. SVC measures the volume that can be exhaled from a full inhalation after exhaling to a maximum as slowly as possible. The percent (%) of predicted SVC is reported.
Time Frame: Week 76 (or end of trial)
Population: modified intention-to-treat (mITT)
Measure: Mean (Standard Deviation); unit: percent (%) predicted SVC
Arm/Group | Arimoclomol (up to 76 Weeks) | Placebo (up to 76 Weeks)
Number analyzed (Participants) | 160 | 79
percent (%) predicted SVC | -30.65 (26.346) | -30.38 (23.839)

ADVERSE EVENTS:
Time Frame: From first dose of study medication up to 76 weeks. Assessed every week.
Description: The safety population included all participants not on edaravone at baseline who received any amount of study medication.
  The safety analysis included all events occurring during the on-treatment observation period which started at the date of first administration of study medication and until 14 days following the latest administration of study medication (in case of interruption of treatment) or last dose of study medication, or end of trial, whichever is earliest.
Arm/Group | Arimoclomol (up to 76 Weeks) | Placebo (up to 76 Weeks)
All-Cause Mortality (participants affected / at risk) | 29/160 | 18/79
Serious Adverse Events (participants affected / at risk) | 36/160 | 20/79
Other Adverse Events (participants affected / at risk) | 149/160 | 71/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arimoclomol (up to 76 Weeks) (N=160) | Placebo (up to 76 Weeks) (N=79)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 5
Respiratory tract infection (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Hepatic enzyme increased (Investigations) | 2 | 0
Transaminases increased (Investigations) | 2 | 0
Medical observation (Investigations) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Oesophageal perforation (Gastrointestinal disorders) | 0 | 1
Medical device site inflammation (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Assisted suicide (Psychiatric disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Pupils unequal (Eye disorders) | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arimoclomol (up to 76 Weeks) (N=160) | Placebo (up to 76 Weeks) (N=79)
Headache (Nervous system disorders) | 34 | 21
Fall (Injury, poisoning and procedural complications) | 33 | 17
Constipation (Gastrointestinal disorders) | 32 | 10
Insomnia (Psychiatric disorders) | 23 | 7
Nausea (Gastrointestinal disorders) | 27 | 3
Nasopharyngitis (Infections and infestations) | 14 | 15
Diarrhoea (Gastrointestinal disorders) | 16 | 8
Pneumonia (Infections and infestations) | 10 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 7
Dizziness (Nervous system disorders) | 16 | 4
Oedema peripheral (General disorders) | 15 | 5
Urinary tract infection (Infections and infestations) | 12 | 7
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 10 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 5
Depression (Psychiatric disorders) | 8 | 7
Influenza (Infections and infestations) | 10 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 5
Contusion (Injury, poisoning and procedural complications) | 9 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 2
Bronchitis (Infections and infestations) | 6 | 5
Alanine aminotransferase increased (Investigations) | 9 | 2
Dyspepsia (Gastrointestinal disorders) | 6 | 5
Fatigue (General disorders) | 9 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 | 4
Rash (Skin and subcutaneous tissue disorders) | 9 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 4
Procedural pain (Injury, poisoning and procedural complications) | 5 | 4
Flatulence (Gastrointestinal disorders) | 4 | 4
Hypertension (Vascular disorders) | 4 | 4
Sleep disorder (Psychiatric disorders) | 3 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT03491462/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT03491462/SAP_001.pdf